CLINICAL TRIAL: NCT01966900
Title: A Phase 1 Open-Labelled Trial to Evaluate the Safety and Immunogenicity of CN54gp140 in HIV-Uninfected, Healthy Volunteers
Brief Title: The Safety and Immunogenicity of a Potential HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: X001
Record Dates: First submitted 2013-10-15; First posted 2013-10-22 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: HIV Infections
Keywords: Human immunodeficiency disease; HIV; Vaccine; CN54gp140; Glucopyranosyl lipid adjuvant; GLA; GLA-AF
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Biological/Vaccine: CN54gp140 mixed with GLA-AF
  Vaccination at Months 0, 1, 2 and 6; each vaccination an intramuscular injection of 100 micrograms CN54gp140 mixed with 5 micrograms GLA-AF
  Interventions: Biological: CN54gp140 mixed with GLA-AF
- Group B (Active Comparator): Biological/Vaccine: CN54gp140 mixed with GLA-AF
  Vaccination at Months 0, 1, 2 and 12; each vaccination an intramuscular injection of 100 micrograms CN54gp140 mixed with 5 micrograms GLA-AF
  Interventions: Biological: CN54gp140 mixed with GLA-AF

INTERVENTIONS:
Biological: CN54gp140 mixed with GLA-AF — Each vaccination an intramuscular injection of 100 micrograms CN54gp140 mixed with 5 micrograms GLA-AF

SUMMARY:
The potential HIV vaccine has two components: a protein immunogen based on the coat protein of HIV; and an adjuvant which enhances the vaccinee's response to the immunogen. The immunogen is CN54gp140, and the adjuvant is glucopyranosyl lipid adjuvant - aqueous formulation (GLA-AF).

We wish to assess the vaccine's safety and immunogenicity (the nature of the immune response stimulated by the vaccine) when it is given in two different dose regimens:

Group A: vaccinations at Months 0, 1, 2 and 6; and Group B: vaccinations at Months 0, 1, 2 and 12.

Each dose will be an intramuscular injection of 100 micrograms of CN54gp140 mixed with 5 micrograms of GLA-AF.

We will recruit only healthy, HIV-uninfected men and women. We will assess the safety of the vaccine by monitoring the occurrence of adverse events in the participants. We will assess the immunogenicity of the vaccine by monitoring the immune response to the vaccine in blood and in genital mucosal secretion samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, as assessed by medical history, physical exam, and laboratory tests;
* At least 18 years of age on the day of screening and has not reached his/her 46th birthday on the day of first vaccination;
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study;
* Willing and able to give written informed consent;
* Willing to undergo HIV testing, receive HIV test results and be committed to maintaining low risk behaviour for the trial duration;
* If a female who is sexually active with male partner(s), willing to use an effective method of contraception from screening until at least 4 months after the last study vaccination [e.g., hormonal contraceptives, consistent record with condoms, physiological or anatomical sterility in self or partner, but excluding intrauterine device (IUD) which would preclude the collection of cervico-vaginal secretions with Softcup];
* All female volunteers must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Procedures (Appendices A-B) and must test negative prior to each study vaccination;
* All sexually active males (unless anatomically sterile or in a monogamous relationship with a female partner who uses a documented non-barrier method of birth control) must be willing to use an effective method of contraception (e.g., consistent condom use) from the day of first vaccination until at least 4 months after the last vaccination;
* Willing to forgo donations of blood or any other tissues during the study and, for those who test HIV-positive due to trial vaccination (vaccine-induced HIV seropositivity), until the anti-HIV antibody titres become undetectable.
* Registered with a general practitioner for at least the past three months

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection;
* Any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted); immunosuppressive, anti-cancer, anti-tuberculosis or other medications considered significant by the investigator within the previous 6 months;
* Any clinically significant acute or chronic medical condition that is considered progressive, or in the opinion of the investigator, makes the volunteer unsuitable for participation in the study;
* Reported risky behaviour for HIV infection within the 6 months prior to vaccination as defined by: history of injecting drug use in the previous ten years; gonorrhoea or syphilis in the last six months; high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months; unprotected anal intercourse in the last six months, outside a relationship with a regular partner known to be HIV negative; or unprotected vaginal intercourse in the last six months outside a relationship with a regular known/presumed HIV negative partner.
* Reported abnormal cervical cytology or previous or ongoing treatment for Cervical Intraepithelial Neoplasia;
* If female, pregnant or planning a pregnancy within 4 months after last study vaccination; or lactating;
* Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions) (Note: A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has intramuscular injections and blood draws without any adverse experience, is eligible);
* History of splenectomy;
* Any of the following abnormal laboratory parameters listed below: haemoglobin <11.0 g/dL; absolute neutrophil count (ANC) ≤ 1.3 x 109/L; absolute lymphocyte count (ALC) ≤ 0.9 x 109/L; platelets ≤ 125 x 109/L; creatinine >1.1 x upper limit of normal (ULN); aspartate aminotransferase >1.25 x ULN; alanine aminotransferase >1.25 x ULN; clinically significant abnormal urinalysis dipstick confirmed by microscopy (protein 2+ or more, blood 2+ or more not due to menses); positive for hepatitis B surface antigen (HbsAg), hepatitis C (HCV antibodies) or active syphilis;
* Receipt of live-attenuated vaccine within the previous 60 days or planned receipt within 60 days after vaccination with Investigational Product; or receipt of other vaccine, allergy treatment with antigen injections or tuberculin skin test within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product;
* Receipt of blood transfusion or blood-derived products within the previous 3 months;
* Participation in another clinical trial of an Investigational Product currently, within the previous 3 months or expected participation during this study;
* Prior receipt of another investigational HIV vaccine candidate (Note: receipt of placebo in a previous HIV vaccine trial will not exclude a volunteer from participation if documentation is available);
* History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulty, angioedema);
* Psychiatric condition that compromises safety of the volunteer and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years;
* Seizure disorder: a participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years.);
* If female, history of toxic shock syndrome (TSS), which would preclude the use of Softcup;
* If female, current use of intrauterine device (IUD), which would preclude the use of Softcup;
* If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fidler, MD, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Anderson J, Olafsdottir TA, Kratochvil S, McKay PF, Ostensson M, Persson J, Shattock RJ, Harandi AM. Molecular Signatures of a TLR4 Agonist-Adjuvanted HIV-1 Vaccine Candidate in Humans. Front Immunol. 2018 Feb 26;9:301. doi: 10.3389/fimmu.2018.00301. eCollection 2018. PMID 29535712
- [Derived] Kratochvil S, McKay PF, Kopycinski JT, Bishop C, Hayes PJ, Muir L, Pinder CL, Cizmeci D, King D, Aldon Y, Wines BD, Hogarth PM, Chung AW, Kent SJ, Held K, Geldmacher C, Dally L, Santos NS, Cole T, Gilmour J, Fidler S, Shattock RJ. A Phase 1 Human Immunodeficiency Virus Vaccine Trial for Cross-Profiling the Kinetics of Serum and Mucosal Antibody Responses to CN54gp140 Modulated by Two Homologous Prime-Boost Vaccine Regimens. Front Immunol. 2017 May 24;8:595. doi: 10.3389/fimmu.2017.00595. eCollection 2017. PMID 28596770

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Biological/Vaccine: CN54gp140 mixed with GLA-AF
  Vaccination at Months 0, 1, 2 and 6; each vaccination an intramuscular injection of 100 micrograms CN54gp140 mixed with 5 micrograms GLA-AF
  CN54gp140 mixed with GLA-AF: Each vaccination an intramuscular injection of 100 micrograms CN54gp140 mixed with 5 micrograms GLA-AF
- Group B: Biological/Vaccine: CN54gp140 mixed with GLA-AF
  Vaccination at Months 0, 1, 2 and 12; each vaccination an intramuscular injection of 100 micrograms CN54gp140 mixed with 5 micrograms GLA-AF
  CN54gp140 mixed with GLA-AF: Each vaccination an intramuscular injection of 100 micrograms CN54gp140 mixed with 5 micrograms GLA-AF
Period: Overall Study
Arm/Group | Group A | Group B
Started | 8 | 6
Completed | 6 | 6
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate or Greater Reactogenicity (i.e., Solicited Adverse Events)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
Participants | 2 | 4

2. Primary Outcome: Number of Participants With Moderate or Greater and/or Vaccine-related Unsolicited Adverse Events (AEs)
Description: Including safety laboratory (biochemical, haematological) parameters, from the day of each vaccination up to 28 days post each vaccination.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
Participants | 3 | 3

3. Primary Outcome: Number of Participants With Vaccine Related Serious Adverse Events (SAEs) Collected Throughout the Study Period
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 months
Description: Data on local and systemic reactogenicity (i.e., solicited adverse events) was collected by structured interview and medical examination at clinic visits. Data on other adverse events was collected with open-ended questions. Volunteers were given diary cards as a memory aid for collecting adverse events during the 7 days after each vaccination.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=8) | Group B (N=6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 2 or higher
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) — Grade 2 or higher
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) — Grade 2 or higher
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2 or higher
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 2 or higher
Headache (Nervous system disorders) | 1 (1) | 2 (2) — Grade 2 or higher
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) — Grade 2 or higher
Myalgia (General disorders) | 2 (2) | 0 (0) — Grade 2 or higher
Malaise (General disorders) | 1 (1) | 3 (3) — Grade 2 or higher
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2 or higher
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2 or higher
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) — Grade 2 or higher

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes